CLINICAL TRIAL: NCT02346656
Title: BRAVO: a BavaRiAn eValuatiOn of DRG Stimulation for the Treatment for Chronic Post Surgical Pain of the Groin
Brief Title: a BavaRiAn eValuatiOn of Dorsal Root Ganglion (DRG) Stimulation for the Treatment for Chronic Post Surgical Pain of the Groin
Acronym: BRAVO
Status: Terminated | Type: Observational
Why Stopped: Inadequate Enrolment
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-SMI-2013
Record Dates: First submitted 2015-01-09; First posted 2015-01-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Post Surgical Groin Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated subjects: All subjects recruited and treated with the Axium neurostimulator
  Interventions: Device: Implantation with the commercially available Axium neurostimulator

INTERVENTIONS:
Device: Implantation with the commercially available Axium neurostimulator

SUMMARY:
15-SMI-2013 is a post market, observational, questionnaire based study to assess the effectiveness of the commercially available Axium neurostimulator in the management of chronic post surgical groin pain

ELIGIBILITY:
Inclusion Criteria:

1. The patient is at least 18 years old
2. The patient is willing and able to comply with the examination schedule and the trial schedule.
3. The patient has suffered from chronic post-surgical neuropathic groin pain for at least 6 months
4. Conservative treatments of the chronic pain including medication, physiotherapy and interventions have been exhausted
5. The pain level at the time of the baseline examination is at least 60mm on the visual analogue scale (VAS) in the primary pain area (groin pain)
6. The patient is able to give consent in writing

Exclusion Criteria:

1. Pregnant or breastfeeding patients or those who plan to become pregnant during the study
2. It has been established in an examination by the tester that the pain has significantly worsened or changed its characteristics in the course of the previous month.
3. In the last 30 days, the patient has been treated with corticosteroids on an area scheduled for the stimulation.
4. In the last 3 months, the patient has been treated with radio frequency therapy on an area scheduled for the stimulation.
5. The patient has already been treated with an active implantable device, including an implantable cardioverter defibrillator, pacemaker, spinal cord stimulator or an intrathecal medication pump.
6. The patient is not able to operate the stimulation device
7. The patient is currently suffering from an infection
8. The patient has participated in another clinical study in the last 30 days
9. The patient has a coagulation disorder or is taking anti-coagulants, which would make participation impossible, as per the study doctor
10. The patient has been diagnosed with a malignancy in the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post Surgical Groin Pain Patients
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pain Relief - Assessed by Change in Pain Intensity Assessed using a Visual Analogue Scale (VAS) from Pre-Treatment Baseline | Post treatment at; 1 week and 1, 3, 6 and12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Algesiologikum Zentrum für Schmerzmedizin, München, Germany